CLINICAL TRIAL: NCT03221907
Title: A Multi-center, Randomized, Double-blind, Parallel, Active-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of 'GLA5PR GLARS-NF1 Tab.' and 'Pregabalin' in Peripheral Neuropathic Pain
Brief Title: Clinical Trial to Evaluate the Efficacy and Safety of 'GLA5PR GLARS-NF1 Tab.' in Peripheral Neuropathic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW1502-301
Record Dates: First submitted 2017-07-11; First posted 2017-07-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Pain of Mononeuropathy
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GLA5PR GLARS-NF1 & Pregabalin placebo (Experimental): GLA5PR GLARS-NF1 150mg, 300mg tablet by mouth, every after dinner for about 3 months Pregabalin placebo 75mg, 150mg, 300mg capsules by mouth, every after breakfast and dinner for about 3 months
  Interventions: Drug: GLA5PR GLARS-NF1; Drug: Pregabalin placebo
- GLA5PR GLARS-NF1 placebo & Pregabalin (Active Comparator): GLA5PR GLARS-NF1 placebo 150mg, 300mg tablet by mouth, every after dinner for about 3 months Pregabalin 75mg, 150mg, 300mg capsules by mouth, every after breakfast and dinner for about 3 months
  Interventions: Drug: GLA5PR GLARS-NF1 placebo; Drug: Pregabalin

INTERVENTIONS:
Drug: GLA5PR GLARS-NF1 — Pregabalin tablet
  Arms: GLA5PR GLARS-NF1 & Pregabalin placebo
Drug: GLA5PR GLARS-NF1 placebo — tablet manufactured to mimic GLA5PR GLARS-NF1
  Other Names: placebo (for GLA5PR GLARS-NF1)
  Arms: GLA5PR GLARS-NF1 placebo & Pregabalin
Drug: Pregabalin — Pregabalin capsule
  Other Names: Lyrica
  Arms: GLA5PR GLARS-NF1 placebo & Pregabalin
Drug: Pregabalin placebo — tablet manufactured to mimic pregabalin capsule
  Other Names: placebo (for pregablin)
  Arms: GLA5PR GLARS-NF1 & Pregabalin placebo

SUMMARY:
A multi-center, randomized, double-blind, parallel, active-controlled phase III clinical trial to evaluate the efficacy and safety of 'GLA5PR GLARS-NF1 Tab.' and 'Pregabalin' in peripheral neuropathic pain

ELIGIBILITY:
Inclusion Criteria:

* both male and female who are over 19-year-old
* patient whose pain scale is 4~9
* patient who has pain of mononeuropathy

Exclusion Criteria:

* patient whose CCr is <60ml/min
* patient who has other pain which is not from mononeuropathy
* patient who is going to have an operation during this study
* patient who has abnormal ECG

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2016-04-11 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Daily Pain Rating Scale | 12-week

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee MK, Jeon Y, Choi SS, Lee PB, Kim YC, Suh JH, Sim SE, Song SO, Ko Y, Yu JM, Min K, Lee JH. Efficacy and Safety of the Controlled-release Pregabalin Tablet (GLA5PR GLARS-NF1) and Immediate-release Pregabalin Capsule for Peripheral Neuropathic Pain: A Multicenter, Randomized, Double-blind, Parallel-group, Active-controlled, Phase III Clinical Trial. Clin Ther. 2020 Dec;42(12):2266-2279. doi: 10.1016/j.clinthera.2020.10.009. Epub 2020 Nov 30. PMID 33272643